CLINICAL TRIAL: NCT00859612
Title: Renal Osteodystrophy: A Fresh Approach
Status: Completed | Type: Observational
Sponsor: Hartmut Malluche, MD (Other)
Responsible Party: Sponsor-Investigator, Hartmut Malluche, MD, Professor and Chief, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 1R01DK080770-01A1 (NIH); 1R01DK080770-01A1 (NIH)
Record Dates: First submitted 2009-03-09; First posted 2009-03-11 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Renal Osteodystrophy
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples and bone biopsy samples
Oversight: Data Monitoring Committee: No

SUMMARY:
There are two major goals of this project:

1. Comparison of DXA and QCT for diagnosis of bone loss in CKD-5 patients and determination of the prevalence of low bone turnover in CKD-5 patients with bone loss.
2. Identification of the optimal combination of noninvasive tests for definition of the turnover component of ROD.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older;
* Chronic maintenance dialysis of at least 3 months' duration;
* Mental competence;
* Willingness to participate in the study;
* Calcidiol levels within normal range.

Exclusion Criteria:

* Pregnancy;
* Systemic illnesses or organ diseases that may affect bone (except type 1 or type 2 diabetes mellitus);
* Clinical condition that may limit study participation (e.g., unstable angina, respiratory distress, infections).
* Chronic alcoholism and/or drug addiction;
* Participation in a study of an investigational drug during the past 90 days;
* Allergy to tetracycline.
* Planning to move out of the area within 2 years of the study;
* On active transplant list;
* Treatment within last 6 months with drugs that may affect bone metabolism (except for treatment with calcitriol, vitamin D analogs and/or calcimimetics).
* Calcidiol level below the normal range. The current routine clinical practice in our dialysis clinics is to check calcidiol status twice yearly and supplement with vitamin D according to serum calcidiol levels. It is therefore unlikely that a substantial number of patients will be excluded due to this exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients from dialysis clinics
Sampling Method: Non-Probability Sample
Enrollment: 464 (Actual)
Dates: Start 2009-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Comparison of DXA and QCT for diagnosis of bone loss in CKD-5 patients and determination of the prevalence of low bone turnover in CKD-5 patients with bone loss. | 4 years
  Because each method (QCT or DXA) yields a dichotomous response (bone loss: yes or no), the proportion of patients with a bone loss will be compared between the 2 methods by using the McNemar statistic for correlated proportions.

SECONDARY OUTCOMES:
Identification of the optimal combination of noninvasive tests for definition of the turnover component of ROD. | 4 years
  A stepwise logistic model will be used to determine which combination of PTH and bone markers best predicts low bone turnover.

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut H Malluche, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States